CLINICAL TRIAL: NCT00284011
Title: Effect of the Dietary Supplement S-Adenosyl-L-Methionine on Plasma Homocysteine Levels in Healthy Human Subjects
Brief Title: Effect of the Dietary Supplement SAMe on Blood Homocysteine Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 677-04
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Heart Disease
Keywords: SAMe; AdoMet; Methylation; Homocysteine; Dietary Supplement; S-Adenosyl-L-Methionine
MeSH Terms: conditions — Heart Diseases | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAMe (Active Comparator): Two 400 mg pills.
  Interventions: Dietary Supplement: SAMe
- Placebo (Placebo Comparator): Two placebo pills (identical in appearance to SAMe).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: SAMe — 800 mg dose daily for 4 weeks.
  Other Names: AdoMet; S-Adenosyl-L-Methionine
  Arms: SAMe
Other: Placebo — 2 placebo pills daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the oral intake of the dietary supplement SAMe increases blood homocysteine levels in healthy human subjects.

DETAILED DESCRIPTION:
S-adenosyl-L-methionine (SAMe or AdoMet) is a commonly used nutritional supplement available in the United States since 1999. SAMe is metabolized to homocysteine, a known cardiovascular risk factor. No study has determined the effect exogenous SAMe administration has on the long-term levels of homocysteine in humans. As a nutritional supplement, SAMe is not regulated by the Food and Drug Administration, despite being used to treat clinical diseases such as depression and osteoarthritis.

ELIGIBILITY:
Inclusion criteria:

* Women and men age 18 - 65
* Able to understand and sign a consent form

Exclusion criteria:

* Smoking
* Pregnant or lactating
* Women actively trying to conceive
* Diagnosis of panic disorder or bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Homocysteine levels pre- and post- one month of SAMe administration. | 1 Month

SECONDARY OUTCOMES:
An interim (2 week) homocysteine level, high sensitivity C-reactive protein (hsCRP) level, lipid studies, and liver blood tests. | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dietland Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Thompson MA, Bauer BA, Loehrer LL, Cha SS, Mandrekar JN, Sood A, Wahner-Roedler DL. Dietary supplement S-adenosyl-L-methionine (AdoMet) effects on plasma homocysteine levels in healthy human subjects: a double-blind, placebo-controlled, randomized clinical trial. J Altern Complement Med. 2009 May;15(5):523-9. doi: 10.1089/acm.2008.0402. PMID 19422296